CLINICAL TRIAL: NCT00509106
Title: A Phase 3, Multicenter, Randomized, Double-blind, Comparative Study to Evaluate the Safety and Efficacy of Ceftaroline Versus Ceftriaxone in the Treatment of Adult Subjects With Community-Acquired Pneumonia
Brief Title: Comparative Study of Ceftaroline vs. Ceftriaxone in Adults With Community-Acquired Pneumonia
Acronym: CAP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P903-09
Record Dates: First submitted 2007-07-27; First posted 2007-07-31 (Estimated); Results first posted 2010-11-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-02

CONDITIONS: Bacterial Pneumonia
Keywords: ceftaroline; Community-acquired pneumonia; CAP; Streptococcus pneumoniae; Haemophilus influenzae; Mycoplasma pneumoniae; Chlamydophila spp; Legionella ssp; multi-drug resistant Streptococcus pneumoniae (MDRSP); antimicrobial resistance; pneumococci; beta-lactam; ceftaroline fosamil; ceftriaxone; antibiotic
MeSH Terms: conditions — Pneumonia, Bacterial; Community-Acquired Pneumonia; Haemophilus Infections | interventions — Ceftaroline; Injections; Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ceftaroline fosamil for injection (Experimental): Ceftaroline fosamil was administered in two consecutive 300 mg IV infusions over 30 minutes, every 12 hours (q12h).
  Interventions: Drug: Ceftaroline fosamil for Injection
- IV Ceftriaxone (Active Comparator): Ceftriaxone was administered as a 1-g IV infusion over 30 minutes followed by IV saline placebo infused over 30 minutes, every 24 hours (q24h).
  Interventions: Drug: Ceftriaxone; Drug: Placebo

INTERVENTIONS:
Drug: Ceftaroline fosamil for Injection — 2 consecutive, 300 mg dose parenteral infused over 30 minutes, every 12 hours for 5 to 7 days
  Other Names: Experimental
  Arms: Ceftaroline fosamil for injection
Drug: Ceftriaxone — 1 g dose parenteral infused over 30 minutes, every 24 hours for 5 to 7 days
  Other Names: Active comparator
  Arms: IV Ceftriaxone
Drug: Placebo — Subjects randomized to receive ceftriaxone will receive ceftriaxone at a dose of 1 g infused over 30 minutes followed by IV saline placebo infused over 30 minutes, every 24 hours (q24h). Twelve hours after each dose of ceftriaxone and saline placebo (ie, between ceftriaxone doses), subjects in this group will receive two consecutive saline placebo infusions, each infused over 30 minutes q24h. The ceftriaxone and saline placebo infusions will correspond to the q12h infusions of ceftaroline, thereby maintaining the blind
  Arms: IV Ceftriaxone

SUMMARY:
The purpose of the study is to determine if the antibiotic ceftaroline is safe and effective in the treatment of community-acquired pneumonia in adults.

DETAILED DESCRIPTION:
Clinical trials is being held in different countries. The purpose of the study is to determine if the antibiotic ceftaroline is safe and effective in the treatment of community-acquired pneumonia in adults.

ELIGIBILITY:
Inclusion Criteria:

Subjects with community-acquired pneumonia requiring:

* initial hospitalization or treatment in an emergency room or urgent care setting
* infection requiring initial treatment with IV antimicrobial

Exclusion Criteria:

* Community-acquired pneumonia suitable for outpatient therapy with an oral antimicrobial agent
* Respiratory tract infections not due to community-acquired bacterial pathogens
* Infections resistant to ceftriaxone
* Any condition requiring concomitant systemic corticosteroids
* History of any hypersensitivity or allergic reaction to any ß-lactam antimicrobial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 622 (Actual)
Dates: Start 2007-07; Primary Completion 2008-08 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: IM Hoepelman, MD, Principal Investigator — UMC Utrecht
Locations (91):
- Investigational Site, Durham, North Carolina, United States
- Argentina (12):
  - Investigational Site, Autonoma, Buenos Aires
  - Investigational Site, Mar del Plata, Buenos Aires
  - Investigational Site, Merlo, Buenos Aires
  - Investigational Site, Córdoba, Córdoba Province
  - Investigational Site, Buenos Aires
  - Invetigational Site, Buenos Aires
  - Investigational Site, Córdoba
  - INvestigational Site, Córdoba
  - Investigational Site, Entre Ríos
  - Investigational Site, Granadero Baiggoria
  - Investigational Site, Paraná
  - Investigational Site, Santa Fe
- Austria (4):
  - Investigational site, Grieskirchner, Wels
  - Investigational Site, Steyr
  - Investigational Site, Vienna
  - Investigational Site, Wels
- Bulgaria (4):
  - Investigational Site, Plovdiv
  - Investigational Site, Rousse
  - Investigational Site, Sofia
  - Investigational Drug, Varna
- Chile (7):
  - Investigational Site, San Ignacio, Región de Valparaíso
  - Investigational Site, Santiago
  - Investigational Site, Talcahuano
  - Investigational Site, Temuco
  - Inestigational Site, Valdivia
  - Investigational Site, Valdivia
  - Investigational Site, Valparaíso
- Germany (15):
  - Investigational Site, Aachen
  - Investigational Site, Berlin
  - Inestigational Site, Berlin
  - Investigational Site, Dachau
  - Investigational Site, Frankfurt
  - Investigational Site, Frankfurt am Main
  - Investigational Site, Greifswald
  - Investigational Site, Halle
  - Investigtional Site, Hanover
  - Investigational Site, Heidelberg
  - Investigational Site, Hofheim
  - Investigational Site, Immenhausen
  - Investigational Site, Lübeck
  - Investigational Site, Rotenburg (Wümme)
  - Investigational Site, Wuppertal
- Hungary (7):
  - Investigational Site, Győr
  - Investigational Site, Nyíregyháza
  - Investigational Site, Seregelyesi
  - Investigational Site, Sostoi
  - Investigational Site, Szent Instvan
  - Investigational Site, Székesfehérvár
  - Investigational Site, Vasvari Pal
- India (5):
  - Investigational Site, Bangalore
  - Investigational Site, Gujarat
  - Investigational Site, Karnataka
  - Investigational Site, Noida
  - Investigational Site, Pradesh
- Latvia (4):
  - Investigational Site, Daugavpils
  - Investigational Site, Latvia
  - Investigational Site, Liepāja
  - Investigational Site, Riga
- Mexico (4):
  - Investigational Site, Chihuahua City
  - Investigational Site, Jalisco
  - Investigational Site, Lima
  - Investigational Site, Sonora
- Investigational Site, Lima, Peru
- Poland (14):
  - Investigator Site, Bialystok
  - Investigational Site, Bystra
  - Investigational Site, Chrzanów
  - Investigational Site, Krakow
  - Investigtional Site, Krakow
  - Investigational Site, Lodz
  - Investigational Site, Lublin
  - Investigational Site, Poznan
  - Investigational Site, Skierniewice
  - Inestigational Site, Warsaw
  - Investigational Site, Warsaw
  - Investigational Site, Wilkowice-Bystra
  - Investigational Site, Wroclaw
  - Investigational Site, Zabrze
- Romania (2):
  - Investigational Site, Bucharest
  - Investigational Site, Craiova
- Russia (4):
  - Investigational Site, Moscow
  - Investigational Site, Saint Petersburg
  - Investigational Site, Smolensk
  - Investigational Site, Yaroslavl
- Ukraine (7):
  - Investigational Site, Dnipropetrovsk
  - Investigational Site, Kharkiv
  - Investigational site, Kyiv
  - Investigational Site, Kyiv
  - Investigational Site, Vinnytsia
  - Investigational Site, Zaporizhya
  - Investigational Site, Zhytomyr

REFERENCES:
- [Derived] Dryden M, Kantecki M, Yan JL, Stone GG, Leister-Tebbe H, Wilcox M. Treatment outcomes of secondary bacteraemia in patients treated with ceftaroline fosamil: pooled results from six phase III clinical trials. J Glob Antimicrob Resist. 2022 Mar;28:108-114. doi: 10.1016/j.jgar.2021.10.027. Epub 2021 Dec 16. PMID 34922058
- [Derived] Cheng K, Pypstra R, Yan JL, Hammond J. Summary of the safety and tolerability of two treatment regimens of ceftaroline fosamil: 600 mg every 8 h versus 600 mg every 12 h. J Antimicrob Chemother. 2019 Apr 1;74(4):1086-1091. doi: 10.1093/jac/dky519. PMID 30597021
- [Derived] Taboada M, Melnick D, Iaconis JP, Sun F, Zhong NS, File TM, Llorens L, Friedland HD, Wilson D. Ceftaroline fosamil versus ceftriaxone for the treatment of community-acquired pneumonia: individual patient data meta-analysis of randomized controlled trials. J Antimicrob Chemother. 2016 Apr;71(4):862-70. doi: 10.1093/jac/dkv415. Epub 2015 Dec 24. PMID 26702925
- [Derived] Lodise TP, Anzueto AR, Weber DJ, Shorr AF, Yang M, Smith A, Zhao Q, Huang X, File TM. Assessment of time to clinical response, a proxy for discharge readiness, among hospitalized patients with community-acquired pneumonia who received either ceftaroline fosamil or ceftriaxone in two phase III FOCUS trials. Antimicrob Agents Chemother. 2015 Feb;59(2):1119-26. doi: 10.1128/AAC.03643-14. Epub 2014 Dec 8. PMID 25487791
- [Derived] Shorr AF, Kollef M, Eckburg PB, Llorens L, Friedland HD. Assessment of ceftaroline fosamil in the treatment of community-acquired bacterial pneumonia due to Streptococcus pneumoniae: insights from two randomized trials. Diagn Microbiol Infect Dis. 2013 Mar;75(3):298-303. doi: 10.1016/j.diagmicrobio.2012.12.002. Epub 2013 Jan 26. PMID 23357290
- [Derived] Rank DR, Friedland HD, Laudano JB. Integrated safety summary of FOCUS 1 and FOCUS 2 trials: Phase III randomized, double-blind studies evaluating ceftaroline fosamil for the treatment of patients with community-acquired pneumonia. J Antimicrob Chemother. 2011 Apr;66 Suppl 3:iii53-9. doi: 10.1093/jac/dkr099. PMID 21482570
- [Derived] Low DE, File TM Jr, Eckburg PB, Talbot GH, David Friedland H, Lee J, Llorens L, Critchley IA, Thye DA; FOCUS 2 investigators. FOCUS 2: a randomized, double-blinded, multicentre, Phase III trial of the efficacy and safety of ceftaroline fosamil versus ceftriaxone in community-acquired pneumonia. J Antimicrob Chemother. 2011 Apr;66 Suppl 3:iii33-44. doi: 10.1093/jac/dkr097. PMID 21482568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited worldwide from July 2007 to August 2008
Pre-assignment Details: Patients were screened for up to 24 hours
Period: Overall Study
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Started | 315 | 307
Completed | 284 | 278
Not Completed | 31 | 29
Not completed — Adverse Event | 3 | 2
Not completed — Noncompliance | 0 | 1
Not completed — At the request of sponsor/investigator | 1 | 2
Not completed — Withdrew consent | 4 | 8
Not completed — Lost to Follow-up | 16 | 10
Not completed — Other | 1 | 0
Not completed — Death | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone | Total
Number analyzed (Participants) | 315 | 307 | 622
Age, Customized [Number; unit: participants]
  <65 years | 183 | 173 | 356
  >=65 years | 132 | 134 | 266
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (17.0) | 60.0 (15.5) | 59.5 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 105 | 231
  Male | 189 | 202 | 391

OUTCOME MEASURES:

1. Primary Outcome: Clinical Cure Rate for Ceftaroline Compared to That for Ceftriaxone at the Test of Cure (TOC) in the Modified Intent to Treat Efficacy (MITTE) Population
Description: Cure:Total resolution of all signs and symptoms of pneumonia (ie,CABP), or improvement to such an extent that further antimicrobial therapy was not necessary
  Failure: Any of the following:
  * Persistence, incomplete clinical resolution, or worsening in signs and symptoms of CABP that required alternative antimicrobial therapy
  * Treatment-limiting adverse event (AE) leading to discontinuation of study drug therapy, when subject required alternative antimicrobial therapy to treat the pneumonia
  * Death wherein pneumonia (ie,CABP) was considered causative
  Indeterminate: Inability to determine an outcome
Time Frame: 8-15 days after last dose of study drug
Population: The MITTE Population consisted of all subjects in the MITT Population (all randomized subjects who received any amount of the study drug) in PORT Risk Class III or IV. The Pneumonia Outcomes Research Team (PORT) scale of CAP severity in which Risk Class I is associated with the lowest risk for mortality and Risk Class V represents the highest risk.
Measure: Number; unit: participants
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Number analyzed (Participants) | 315 | 307
participants
  Clinical cure | 235 | 206
  Clinical failure | 47 | 56
  Indeterminate | 7 | 11
Statistical Analysis 1: Comparison: Ceftaroline Fosamil for Injection vs IV Ceftriaxone; The primary objective of this study was to determine the noninferiority in the clinical cure rate for ceftaroline compared with that for ceftriaxone at TOC in the MITTE Population in adult subjects with CABP; Test type: Non-Inferiority or Equivalence — A two-sided 95% Confidence Interval (CI) for the observed difference in the primary outcome measure (clinical cure rate) between the ceftaroline group and the ceftriaxone group was calculated based on the MITTE Population at the TOC visit. Noninferiority was concluded if the lower limit of the 95% CI was higher than -10% for the MITTE populations; Risk Difference (RD) = 5.9, 95% CI 2-sided [-1.0 to 12.7] — Risk difference corresponds to Ceftaroline clinical cure rate minus Ceftriaxone clinical cure rate. The confidence interval was calculated using the Miettinen and Nurminen method without adjustment

2. Primary Outcome: Clinical Cure Rate for Ceftaroline Compared With That for Ceftriaxone at TOC in the Clinically Evaluable (CE) Population
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

3. Secondary Outcome: Clinical Response at End of Therapy (EOT)
Time Frame: Last day of study drug administration
Reporting Status: Not Posted

4. Secondary Outcome: Microbiological Success Rate at TOC
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

5. Secondary Outcome: Overall Clinical and Radiographic Success Rate at TOC
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

6. Secondary Outcome: Clinical and Microbiological Response by Pathogen at TOC
Time Frame: 8-15 days after last dose of study drug
Reporting Status: Not Posted

7. Secondary Outcome: Clinical Relapse at Late Follow Up (LFU) Visit
Time Frame: 21-35 days after last dose of study drug
Reporting Status: Not Posted

8. Secondary Outcome: Microbiological Reinfection/Recurrence at LFU
Time Frame: 21 to 35 days after last dose of study drug
Reporting Status: Not Posted

9. Secondary Outcome: Evaluate Safety
Time Frame: first dose, throughout the treatment period, and up to the TOC visit
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: All safety analysis was performed on the Safety Population, those subjects that had received any amount of actual study drug
Arm/Group | Ceftaroline Fosamil for Injection | IV Ceftriaxone
Serious Adverse Events (participants affected / at risk) | 41/315 | 39/307
Other Adverse Events (participants affected / at risk) | 67/315 | 49/307
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=315) | IV Ceftriaxone (N=307)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Postinfarction angina (Cardiac disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 7 (7) | 4 (4)
Pyothorax (Infections and infestations) | 3 (3) | 0 (0)
Lung abscess (Infections and infestations) | 2 (2) | 3 (3)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis C (Infections and infestations) | 0 (0) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bactgeraemia (Infections and infestations) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Anoxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiovascular insufficiency (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ceftaroline Fosamil for Injection (N=315) | IV Ceftriaxone (N=307)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 9 (9)
Nausea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Hypokalemia (Metabolism and nutrition disorders) | 10 (10) | 5 (5)
Headache (Nervous system disorders) | 11 (11) | 5 (5)
Insomnia (Psychiatric disorders) | 10 (10) | 8 (8)
Hypertension (Vascular disorders) | 8 (8) | 8 (8)
Phlebitis (Vascular disorders) | 10 (10) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No